CLINICAL TRIAL: NCT03098277
Title: Accelerometry to Optimize and Monitor Human Performance in Cancer Chemotherapy Outpatients
Brief Title: Movement Tracking Devices to Monitor Physical Activity in Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0S-16-2; NCI-2016-00627 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-16-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2017-03-31 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Solid Neoplasm
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational (physical activity, PROs) (Experimental): Patients perform 2 physical activities in an exam room that are recorded using a Microsoft Kinect 2 stationary movement tracking device on days 1 and 21. The first activity is rising from a chair, walking 10 feet, and returning to the chair. The second activity is moving from the chair to the step-up examination table. Patients also wear a movement tracking wristband, Microsoft Band 2, around their wrist, complete a smartphone application based PRO questionnaire, and weigh themselves daily for 60 days.
  Interventions: Other: Accelerometer; Other: Laboratory Biomarker Analysis; Other: Physical Activity Measurement; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Accelerometer — Wear Microsoft Band 2
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Physical Activity Measurement — Perform physical activities recorded by Microsoft Kinect 2
  Other Names: ACTIVITY
Behavioral: Telephone-Based Intervention — Complete PRO questionnaires

SUMMARY:
This clinical trial studies movement tracking devices in optimizing and monitoring physical activity in patients with solid tumors undergoing chemotherapy in a health care facility during the day without spending the night. Movement tracking devices, such as Microsoft Kinect 2 and Microsoft Band 2, may help doctors learn about the health of cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of monitoring cancer patients using wrist-worn activity monitors and movement trackers.

SECONDARY OBJECTIVES:

I. To evaluate the association between activity and patient reported fatigue. II. To evaluate the association between movement and incidents of health care interventions (hospitalizations, physical visits, intravenous hydration, etc.)

TERTIARY OBJECTIVES:

I. To compare physician and patient assessed Eastern Cooperative Oncology Group (ECOG) and Karnofsky performance status scores with the data obtained from movement trackers.

OUTLINE:

Patients perform 2 physical activities in an exam room that are recorded using a Microsoft Kinect 2 stationary movement tracking device on days 1 and 21. The first activity is rising from a chair, walking 10 feet, and returning to the chair. The second activity is moving from the chair to the step-up examination table. Patients also wear a movement tracking wristband, Microsoft Band 2, around their wrist, complete a smartphone application based patient reported outcome (PRO) questionnaire, and weigh themselves daily for 60 days.

After completion of study, patients are followed up at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of a solid tumor, undergoing palliative or adjuvant therapy
* Undergoing at least 2 planned cycles of highly emetogenic chemotherapy defined according to the Hekseth scale; the cycles may range in duration from 14 days to 28 days, according to standard of care practices
* Ability to understand and the willingness to sign a written informed consent
* Willingness to wear sensors to track physical activity, Global Positioning System (GPS) location, and provide symptom ratings each night for up to 60 days
* Able to read English, Spanish, or Traditional Mandarin to complete patient reported outcomes
* Able to ambulate without an assistive device
* Able to operate a smartphone and wearable wristband

Exclusion Criteria:

* Patients may not be missing limbs
* Patient does not have a diagnosis of a hematologic malignancy
* Patients with symptomatic brain metastases are excluded from this clinical trial; those with asymptomatic brain metastasis are permitted; it is permissible to have the patient on corticosteroids to eliminate symptoms of brain metastasis
* Patient with a known movement disorder such as Parkinson's disease, choreoathetoid movement disorders, essential tremor if that movement disorder is of sufficient severity to require drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients whose wearable activity monitor provides movement data | Up to 60 days
Percent of patients who achieve "data capture success" defined as having both PRO data and accelerometry data transmitted to the investigators in 80% of the observation days | Up to 60 days
  Patients who are unable to comply and have data transmitted, including technical failures, personal decision, hospitalization, or any other reason are counted as "data capture failures". Data from patients who die while on study will not be replaced but will be included prior to their date of death, days between death and day 60 will not be included in the denominator when calculating "data capture success" rates.

SECONDARY OUTCOMES:
Change in weight over time | Baseline to 60 days
  The relationship between the change in weight over time and patient activity

OTHER OUTCOMES:
Patient in-office activity performance time assessed by Microsoft Kinect 2 | Up to 60 days
  The association between the "get up and go" time and moving onto the examination table will be explored.
Presence of circulating tumor cells in blood | Day 21 (visit 2)
  The association between the presence of circulating tumor cells and patient activity will be explored.
Sum of inpatient and outpatient hospital encounters | Up to 90 days after study discontinuation
  The association between patient movement and the sum of inpatient and outpatient hospital encounters up to 90 days after study discontinuation will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Nieva, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California